CLINICAL TRIAL: NCT00883467
Title: The Effects of Preconditioning on Intramuscular High-Energy Phosphate Levels During Ischemia
Acronym: IPC in MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Prof. Dr. Michael Wolzt, Medical University of Vienna, Department of Clinical Pharmacology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IPC in MRI 040908
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Ischemia
Keywords: Ischemic Preconditioning; functional MRI; BOLD; Reperfusion
MeSH Terms: conditions — Ischemia

ARMS (4):
- 1 (Other): baseline MR signal prior to, during and 30 minutes after an ischemic period of 20 minutes
  Interventions: Procedure: no preconditioning
- 2 (Other): baseline MR signal prior to, during and 30 minutes after an ischemic period of 20 minutes with additional 5 minutes of cuff stenosis directly after cuff release
  Interventions: Procedure: no preconditioning
- 3 (Other): short time preconditioning, other details according arm 2
  Interventions: Procedure: preconditioning
- 4 (Other): long time preconditioning, other details according arm 2
  Interventions: Procedure: preconditioning

INTERVENTIONS:
Procedure: preconditioning — 3 times of five minutes ischemia, produced by cuff inflation to a suprasystolic pressure positioned on the thigh
  Arms: 3; 4
Procedure: no preconditioning — no preconditioning
  Arms: 1; 2

SUMMARY:
Ischemia reperfusion injury may be reduced by ischemic preconditioning. This projects aims to show the effects of short and long time ischemic preconditioning (both sequences 3 x 5 minutes) during and after an ischemic period of 20 minutes in healthy subjects by functional MRI. Ischemia is produces by cuff inflation to a suprasystolic pressure on one tight. Signal is acquired from calf muscles.

A cross-over design of 4 to 8 study periods is used, 4 different study days with 2 different MR measurement methods (BOLD imaging and high energy phosphates) are planned.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 45 years
* Nonsmoker for more than 3 months
* Body mass index between 18 and 25 kg/m2
* Normal findings in medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Evidence of hypertension, pathologic hyperglycemia, hyperlipidemia
* Treatment in the previous 3 weeks with any drug including over-the-counter drugs
* Symptoms of a clinically relevant illness in the 2 weeks before the first study day
* Blood donation during the previous 3 weeks
* Any metallic, electric, electronic or magnetic device or object not removable
* Claustrophobia

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Change in cellular high energy phosphate levels and venous pH concentration for 31P MRS | during and 30 min after ischemia
Main outcome variables: Change in cellular oxygen saturation for BOLD MRI | during and 30 minutes after ischemia
Serum markers of myocellular injury (myoglobin, creatine-kinase) | prior to, directly and 24 hours after ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — MUV, Department of Clinical Pharmacology
Locations (1):
- Medical University of Vienna, Department of Clinical Pharmacology, Vienna, Austria

REFERENCES:
- [Derived] Andreas M, Schmid AI, Keilani M, Doberer D, Bartko J, Crevenna R, Moser E, Wolzt M. Effect of ischemic preconditioning in skeletal muscle measured by functional magnetic resonance imaging and spectroscopy: a randomized crossover trial. J Cardiovasc Magn Reson. 2011 Jun 30;13(1):32. doi: 10.1186/1532-429X-13-32. PMID 21718491